CLINICAL TRIAL: NCT06669559
Title: DROM Test, a Clinical Decision Support Tool for Assessing the Ability to Decide on Returning Home in Elderly Patients with Cognitive Impairments
Brief Title: A Clinical Decision Support Tool for Assessing the Ability to Decide on Returning Home in Elderly Patients with Cognitive Impairments
Acronym: DROM-test
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP240159; 2024-A01838-39 (Other: IDRCB)
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: The Patient's Ability to Decide to Return Home After Hospitalization
Keywords: decision making capacity; dementia; to return home; elderly; capacity assessment
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Person aged 70 and over with a neurocognitive disorder and hospitalized in geriatrics (Other)
  Interventions: Other: DROM-Test

INTERVENTIONS:
Other: DROM-Test — DROM test: a tool for assessing the ability to decide on returning home

SUMMARY:
No validated and generalized tool for assessing a patient's ability to decide whether to return home after hospitalization exists. Evaluating the capacity of elderly patients to decide on their own return home is a daily concern for geriatricians. Neurocognitive disorders do not necessarily mean an inability to decide and the MMSE (mini mental state examination), a reference scale for screening neurocognitive disorders, is not sufficient to determine decision-making capacity apart from extreme scores. Depending on the stage or type of neurocognitive disorders, the same stages of the decision-making process (understanding, reasoning, appreciation, choice) are not impacted. The ability to decide depends on the type of decision (deciding to vote, deciding to take a medication, to participate in clinical research, etc.), i.e. domain-dependent. Associating the clinician's clinical decision with a standardized tool for assessing patients' capacity to decide would enable more ethical clinical practice.

the aim of the study is to add to the clinical decision a decision support tool to assess the capacity to decide whether to return home has better sensitivity in the assessment of the capacity to decide than that of clinical assessment alone

DETAILED DESCRIPTION:
To date, there is no curative treatment for neuro-progressive diseases and it has been shown that cognitive assessment tests such as the MMSE (mini mental state examination) are not sufficient to assess the ability to decide a patient with a neurocognitive disorder.

Evaluating the capacity of elderly patients to decide on their own return home is a daily concern for geriatricians. Indeed, patients with neurocognitive disorders are often forced to be institutionalized without anyone being certain of their inability to decide. 43% of people hospitalized for a short geriatric stay have a neurocognitive disorder linked to Alzheimer's disease. Despite these disorders, it is absolutely necessary to respect the fundamental ethical principles of medical practice and thus the autonomy of the patient. The legal capacity and choice of place of life by the person with or without a disability are protected by international institutions (United Nations (UN), Convention on the Rights of Persons with Disabilities, article 19) and regulated by law, even for patients under legal protection. Neurocognitive disorders do not necessarily mean an inability to decide and the MMSE, the reference scale for screening neurocognitive disorders, is not sufficient to determine decision-making capacity apart from extreme scores. Depending on the stage or type of neurocognitive disorders, the same stages of the decision-making process (understanding, reasoning, appreciation, choice) are not impacted.

The ability to decide depends on the type of decision (deciding to vote, deciding to take medication, participating in clinical research, etc.) or domain-dependent. Currently, the assessment of the ability to decide to return home is carried out by clinicians according to clinical assessment without a specific standardized tool. The variability between evaluators turns out to be very important, specifically identified in the process of being able to decide to take a treatment. Associating the clinician's clinical decision with a standardized tool for evaluating patients' capacity to decide allows for more ethical clinical practice.

No validated and generalized tool for assessing the patient's ability to decide whether to return home after hospitalization exists.

Following this observation, the DROM-test tool (DReam of hOMe), developed within the neuro-psychogeriatrics department of Bretonneau Hospital (102 patients, average age 83 years, average MMSE of 20) allowed to objectify the choice dimension among these four dimensions (understanding, reasoning, appreciation, choice). The performance of the DROM test must now be evaluated on a multicenter scale using an independent expert as the gold standard.

The objective is not to replace the clinical decision but to provide a tool allowing the clinician in his daily practice to argue the decision-making capacity and thus improve the care pathway by increasing the rate of agreement between the clinician and the patient. Failure to return home is often felt as an injustice by patients, providing support for understanding their situation can improve the experience of the situation.

Adding a decision support tool to the clinical decision to assess the capacity to decide whether to return home has better sensitivity in the assessment of the capacity to decide than that of clinical assessment alone.

The population to be studied will be made up of patients with a moderate neurocognitive disorder, a population for which the question of the ability to decide frequently arises, particularly when the patient still lives at home and is weakened by hospitalization. The question of returning home is essential for these patients for whom being sent to a retirement home is experienced as an injustice because it is a non-choice, sometimes even without having been consulted.

The DROM test: The elements of the DROM-test are detailed in the reference publication: 8 questions (understanding, appreciation, choice dimensions) and 4 clinical vignettes (reasoning, choice dimensions) each comprising 3 questions with a binary response.

Its structure includes a questionnaire part and a clinical vignette part improving patients' understanding. Its hetero-questionnaire format, its short administration time (10 min) and its simple instructions make it a tool that could be easily distributed in services receiving elderly people with neurocognitive disorders.

It was improved by taking into account the results of the initial study then after modification, it will be tested on 10 patients from the neuropsychogeriatrics department of Bretonneau hospital in order to reassess the good understanding and consistency of the test.

The DROM-test is given to the patient by their referring doctor. The detailed medical certificate of non-return home: It is a medical certificate produced by an expert doctor registered with a judicial court in France which aims to medically evaluate the capacity of a patient to return home. Usually this certificate is produced for protected adults and sent to the guardianship judge who subsequently decides on any act of disposition of the accommodation.

In this study, it is considered the Gold Standard because the only legally accepted document for this type of evaluation. It will be produced but not sent to court.

ELIGIBILITY:
Inclusion criteria:

* 70 years and over
* neurocognitive disorders regardless of diagnosis
* MMSE between 15 and 25
* hospitalized in geriatrics
* still living at home at the time of hospitalization
* affiliated to or beneficiary of a social security scheme

Non-inclusion criteria

* confusional episode,
* palliative care,
* presence of another significant or systemic pathology: Cerebral Vascular Accident < 3 months, oncological pathology during treatment, decompensated psychiatric illness, acute organ failure,
* total visual or hearing deficit,
* has already taken the DROM test during a previous hospitalization,
* language barrier,
* refusal of participation by the patient, their relative or guardian if applicable
* patient under judicial protection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the DROM test | 3 days
  Ability of the DROM test to accurately identify true positives, meaning patients who truly have the capacity to decide on returning home, according to the gold standard

SECONDARY OUTCOMES:
Specificity of the DROM test | 3 days
  Ability of the DROM test to accurately identify true negatives.
Kappa coefficient of agreement between the initial judgment of the referring physician and their judgment after reviewing the patient's results from the DROM test | 3 days
Percentage of agreement between the clinician and the patient before DROM test | 3 days
Percentage of agreement between the clinician and the patient after DROM test | 3 days
Percentage of patients who completed the DROM test among those who are eligible | 1 year
Percentage of test adherence by patients | 1 year
Percentage of patients who complete the test. | 1 year
Average test duration in minutes | 1 year
Clinician's perception evaluation with the use of the DROM test using a 4-question, 5-point Likert scale (from completely useful to completely useless) | 1 year
Patient's perception evaluation using a 4-question, 5-point Likert scale | 1 year
Description of the factors associated with patients not returning home | 1 year
Optimal DROM-test threshold to identify patients most likely to demonstrate decisional incapacity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mouna Romdhani, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bretonneau, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided